CLINICAL TRIAL: NCT03393793
Title: Heart Transplantation Registry of Pitié-Salpétrière University Hospital
Brief Title: HEart trAnsplantation Registry of piTie-Salpetriere University Hospital
Acronym: HEARTS
Status: Completed | Type: Observational
Sponsor: Lee S Nguyen (Other)
Responsible Party: Sponsor-Investigator, Lee S Nguyen, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Other Study IDs: CIC1421-18-01
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Transplant Disorder; Cardiac Death; Heart Failure; Acute Cellular Graft Rejection; Antibody-Mediated Graft Rejection; Cardiac Allograft Vasculopathy; Heart Transplant Rejection; Immune Tolerance
Keywords: Heart transplantation
MeSH Terms: conditions — Death; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart transplantation (HTx) is a procedure which is hindered by several complications. The HEARTS registry aims to allow the analysis of risk factors of all post-HTx complications. It consists in an exhaustive data collection at the moment of inclusion, i.e. HTx, knowing that patients underwent a full-fledged evaluation beforehand to evaluate their aptitude to being transplanted.

Post-HTx complications include but is not limited to: all-cause mortality, AMR, ACR, CAV, AKI, sepsis, cancer, psychological disorders, metabolic disorders.

DETAILED DESCRIPTION:
Heart transplantation (HTx) is a procedure which is hindered by several complications. The HEARTS registry aims to allow the analysis of risk factors of all post-HTx complications. It consists in an exhaustive data collection at the moment of inclusion, i.e. HTx, knowing that patients underwent a full-fledged evaluation beforehand to evaluate their aptitude to being transplanted.

Post-HTx complications include but is not limited to: all-cause mortality, AMR, ACR, CAV, AKI, sepsis, cancer, psychological disorders, metabolic disorders.

To do so, patients are routinely monitored several times per year, the frequency of which depends on the proximity to the HTx.

An endomyocardial biopsy is performed 3 times per month starting on day 15 until day 65 after HTx, then once every 20 days until four months, then monthly until six months, then once every 45 days until year 1, and every 3 months thereafter until year 2. Afterwards, they become twice per year until year 5, then once a year.

An echocardiography is performed for every visit, with a complete blood analysis, including HLA antibodies screening with DSA evaluation, virologic evaluation.

A coronarography is performed for the anniversary year of HTx, then once every 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplantation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent heart transplantation were included in this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | up to five years after inclusion
  all-cause mortality
Acute cellular rejection (ACR) | up to five years after inclusion
  ACR, biopsy-proven
Antibody mediated rejection (AMR) | up to five years after inclusion
  AMR, biopsy-proven
Acute kidney injury (AKI) | up to five years after inclusion
  AKI, defined by a KDIGO criteria
Severe sepsis or septic shock | up to five years after inclusion
  As defined by Surviving Sepsis Campaign
Cardiac allograft vasculopathy (CAV) | up to five years after inclusion
  CAV, defined ISHLT

CONTACTS AND LOCATIONS:
Overall Officials: Shaida Varnous, MD, Study Director — AP-HP, Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meng P, Nguyen LS, Jabbour F, Ogna A, Clair B, Orlikowski D, Annane D, Lofaso F, Fayssoil A. Accuracy of B-natriuretic peptide for the diagnosis of decompensated heart failure in muscular dystrophies patients with chronic respiratory failure. Neurol Int. 2018 Dec 20;10(4):7917. doi: 10.4081/ni.2018.7917. eCollection 2018 Dec 5. PMID 30687469
- [Result] Nguyen LS, Coutance G, Salem JE, Ouldamar S, Lebreton G, Combes A, Amour J, Laali M, Leprince P, Varnous S. Effect of recipient gender and donor-specific antibodies on antibody-mediated rejection after heart transplantation. Am J Transplant. 2019 Apr;19(4):1160-1167. doi: 10.1111/ajt.15133. Epub 2018 Oct 29. PMID 30286278